CLINICAL TRIAL: NCT00080132
Title: An Open-Label, Dose-Escalating Efficacy and Safety Study of Implitapide in Patients With Hypertriglyceridemia (HTG) on Maximal, Concurrent Triglyceride-Lowering Therapy
Brief Title: Implitapide in Patients With Hypertriglyceridemia (HTG) on Maximal, Concurrent Triglyceride-Lowering Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Medical Research Laboratories International (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: MRL 2002-003
Record Dates: First submitted 2004-03-23; First posted 2004-03-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-04

CONDITIONS: Hypertriglyceridemia
Keywords: HTG; Hypertriglyceridemia, Fredrickson Type I; Hypertriglyceridemia, Fredrickson Type V
MeSH Terms: conditions — Hypertriglyceridemia | interventions — implitapide

INTERVENTIONS:
Drug: implitapide

SUMMARY:
The purpose of this study is to determine if implitapide is effective in lowering triglyceride (TG) levels in patients with Fredrickson Type I or V hypertriglyceridemia where the maximum tolerable medication and diet were not sufficient.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in this study, patients must meet all of the following inclusion criteria:

* be between 8 and 70 years old with diagnosis of Fredrickson Type I or V HTG
* be stable on current maximum tolerated triglyceride lowering therapy
* have a fasting TG level of at least 880 mg/dL (10 mmol/L)
* be male or nonpregnant, nonbreastfeeding female. The women in the study must be surgically sterile, postmenopausal or must practice an effective method of birth control
* must be able to give informed consent or if under the age of 18, parents or legal guardians must give their informed consent
* meet body weight requirements

Exclusion Criteria:

* Recent heart attack, coronary artery intervention, coronary bypass surgery, or stroke.
* Patients with class 3 or 4 heart failure
* Uncontrolled hypothyroidism or other uncontrolled endocrine disease
* Known, clinically significant eye abnormalities, such as cataracts
* History of hepatic disease or AST or ALT levels greater than 1.5 x ULN at Visit 1
* Alkaline phosphatase greater than 2 times ULN
* Serum creatinine greater than 2.0 mg/dL
* Liver cirrhosis and severe liver steatosis
* Clinically significant infection, malignancy, or psychosis
* Use of oral anticoagulants or digoxin unless the dose is stable and is regularly monitored
* Participation in any other investigational study within the last 30 days
* Breastfeeding or pregnant
* Current drug or alcohol abuse
* Serious or unstable medical conditions that would compromise the patient's safety or successful participation in the study
* Unwillingness to comply with study procedures or unwillingness to cooperate fully

Ages: 8 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2004-10; Study Completion 2005-04

CONTACTS AND LOCATIONS:
Locations (9):
- United States (2):
  - Metabolic and Atherosclerosis Research Center, Cincinnati, Ohio
  - The Methodist Hospital, Houston, Texas
- Netherlands (6):
  - Academic Medical Center Amsterdam, Amsterdam
  - Andromed Noord, Groningen
  - Andromed Leiden, Leiden
  - Andromed Rotterdam, Rotterdam
  - Andromed Oost, Velp
  - Andromed Zoetermeer, Zoetermeer
- Lipidklinikken - Rikshospitalet, Oslo, Norway